CLINICAL TRIAL: NCT02412423
Title: Post-transplantation Cyclophosphamide for Haploidentical Transplant From Maternal or Collateral Donors
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiaojun Huang,MD, director, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2015PHB016-01
Record Dates: First submitted 2015-04-05; First posted 2015-04-09 (Estimated); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Hematopoietic Stem Cell Transplantation

ARMS (1):
- treatment group (Experimental): post-transplantation cyclophosphamide
  Interventions: Drug: post-transplantation cyclophosphamide

INTERVENTIONS:
Drug: post-transplantation cyclophosphamide

SUMMARY:
In "beijing model" for haploidentical transplant, the rate of acute graft-versus-host disease (GVHD) from maternal or collateral donors was significantly higher than that from other kins. To reduce the GVHD incidence from maternal or collateral donors, post-transplantation cyclophosphamide is planned to be added into the protocol in "beijing model".

ELIGIBILITY:
Inclusion Criteria:

* haploidentical patients from maternal or collateral donors

Exclusion Criteria:

* uncontrolled infection before transplant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-03; Primary Completion 2016-08 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
rate of acute GVHD | participants will be followed for an expected average of 365 days

SECONDARY OUTCOMES:
rate of non-relapse mortality | participants will be followed for an expected average of 365 days
rate of relapse | participants will be followed for an expected average of 365 days
probability of survival | participants will be followed for an expected average of 365 days

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, China

REFERENCES:
- [Derived] Wang Y, Wu DP, Liu QF, Xu LP, Liu KY, Zhang XH, Yu WJ, Xu Y, Huang F, Huang XJ. Low-dose post-transplant cyclophosphamide and anti-thymocyte globulin as an effective strategy for GVHD prevention in haploidentical patients. J Hematol Oncol. 2019 Sep 3;12(1):88. doi: 10.1186/s13045-019-0781-y. PMID 31481121